CLINICAL TRIAL: NCT04060342
Title: A Phase 1/2, First-in-Human, Open-label, Dose Escalation Study of GB1275 Monotherapy and in Combination With an Anti-PD-1 Antibody in Patients With Specified Advanced Solid Tumors or in Combination With Standard of Care in Patients With Metastatic Pancreatic Adenocarcinoma, Followed by Basket Expansion of GB1275 With Standard of Care or in Combination With an Anti-PD-1 Antibody in Patients With Specified Metastatic Solid Tumors
Brief Title: GB1275 Monotherapy and in Combination With an Anti-PD1 Antibody in Patients With Specified Advanced Solid Tumors or in Combination With Standard of Care in Patients With Metastatic Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No clear benefit of GB1275 was observed either as monotherapy or in combination with pembrolizumab.
Sponsor: GB006, Inc., a wholly owned subsidiary of Gossamer Bio, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Gossamer Bio Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GB1275-1101 (KEYNOTE-A36)
Record Dates: First submitted 2019-08-09; First posted 2019-08-19 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Pancreatic Adenocarcinoma; Esophageal Adenocarcinoma; Esophageal Squamous Cell Carcinoma; Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Triple Negative Breast Cancer; Castration-resistant Prostate Cancer; Microsatellite Stable Colorectal Cancer; Non-small Cell Lung Cancer; Small-cell Lung Cancer; Head and Neck Squamous Cell Carcinoma; Urothelial Carcinoma; Renal Cell Carcinoma; Hepatocellular Carcinoma
Keywords: GEJ adenocarcinoma; TNBC; MSS mCRC; PD-L1 + gastric cancer; PD-L1 positive gastric cancer; NSCLC; SCLC; newly diagnosed stage IV pancreatic adenocarcinoma; HCC; RCC; HNSCC; Transitional Cell Carcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Triple Negative Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Carcinoma, Hepatocellular; Stomach Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Albumin-Bound Paclitaxel; pembrolizumab; spartalizumab

STUDY DESIGN:
Intervention Model Description: Phase 1 - Dose Escalation of 3 different Regimens and Expansion, Phase 2 - Basket Expansion of 3 Cohorts
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Phase 1: Regimen A - GB1275 monotherapy (Experimental): GB1275 Monotherapy dose escalation: Oral administration. Twice per day (BID).
  Interventions: Drug: GB1275
- Phase 1: Regimen B - GB1275 with an Anti-PD-1 (Experimental): GB1275 with pembrolizumab dose escalation and expansion:
  GB1275 oral administration; twice per day (BID), and pembrolizumab IV administration once every 3 weeks (Q3W).
  Interventions: Drug: GB1275; Drug: pembrolizumab
- Phase 1: Regimen C - GB1275 with Standard of Care (SOC) (Experimental): GB1275 with SOC dose escalation:
  GB1275 oral administration; twice per day (BID), and nab-paclitaxel and gemcitabine per United States Prescribing Information (USPI)
  Interventions: Drug: GB1275; Drug: nab-paclitaxel and gemcitabine
- Phase 2: Cohort 1 - GB1275 with SOC (Experimental): GB1275 with SOC Basket Cohort in patients with newly diagnosed metastatic pancreatic cancer:
  GB1275 oral administration; twice per day (BID) and nab-paclitaxel and gemcitabine per USPI.
  Interventions: Drug: GB1275; Drug: nab-paclitaxel and gemcitabine
- Phase 2: Cohort 2 - GB1275 with an Anti-PD-1 (Experimental): GB1275 with pembrolizumab Basket Cohort in patients with MSS colorectal cancer:
  GB1275 oral administration; twice per day (BID), and pembrolizumab IV administration once every 3 weeks (Q3W).
  Interventions: Drug: GB1275; Drug: pembrolizumab
- Phase 2: Cohort 3 - GB1275 with an Anti-PD-1 (Experimental): GB1275 with pembrolizumab Basket Cohort in patients with gastric/GEJ cancer, PD-L1 positive:
  GB1275 oral administration; twice per day (BID), and pembrolizumab IV administration once every 3 weeks (Q3W).
  Interventions: Drug: GB1275; Drug: pembrolizumab

INTERVENTIONS:
Drug: GB1275 — Oral
  Other Names: Investigational
Drug: nab-paclitaxel and gemcitabine — IV infusion
  Other Names: Abraxane and Gemzar
  Arms: Phase 1: Regimen C - GB1275 with Standard of Care (SOC); Phase 2: Cohort 1 - GB1275 with SOC
Drug: pembrolizumab — IV infusion
  Other Names: Anti-PD-1
  Arms: Phase 1: Regimen B - GB1275 with an Anti-PD-1; Phase 2: Cohort 2 - GB1275 with an Anti-PD-1; Phase 2: Cohort 3 - GB1275 with an Anti-PD-1

SUMMARY:
This first-in-human (FIH ) study is an open-label, multicenter study that consists of a Phase 1 Dose Escalation/Expansion phase of GB1275 monotherapy or in combination with Anti-PD-1 Antibody or in combination with Standard of Care in Patients with Metastatic Pancreatic Adenocarcinoma followed by a Phase 2 Basket Expansion phase in Patients with Specified Metastatic Solid Tumors

DETAILED DESCRIPTION:
Note: The Phase 2 portion of the study was not initiated.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* Women of childbearing potential must use an acceptable method of contraception

Phase 1

Subjects with the the following:

* Regimen A and B:

  * pancreatic adenocarcinoma,
  * esophageal adenocarcinoma, or esophageal squamous cell carcinoma, or
  * gastric/gastroesophageal junction adenocarcinoma, or
  * TNBC, or
  * prostate cancer, or
  * colorectal adenocarcinoma, or subjects with tumor types that have progressed after receiving initial treatment benefit rom the last single agent checkpoint inhibitor that is approved for the indication or in combination with standard of care therapy, for example, non-small cell lung cancer, small cell lung cancer, head and neck squamous cell carcinoma, urothelial carcinoma, renal cell carcinoma, and hepatocellular carcinoma, etc.
* Regimen C: newly diagnosed stage IV pancreatic cancer

Phase 2

* Cohort 1: pancreatic cancer.
* Cohort 2: colorectal cancer
* Cohort 3: gastric/GEJ adenocarcinoma

Exclusion Criteria:

* History of another malignancy within 2 years prior to first study drug(s) administration, unless the malignancy was treated with curative intent and the likelihood of relapse is <5% in 2 years
* Pregnant or nursing
* Known history of testing positive for human immunodeficiency virus (HIV)
* Gastrointestinal (GI) tract disease causing the inability to take oral medication.
* Positive test for Hepatitis B virus surface antigen (HBsAg) or a and/or positive Hep C antibody result with detectable hepatitis C virus (HCV) ribonucleic acid (RNA) indicating acute or chronic infection.

Other protocol-defined inclusion/exclusion criteria will apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2022-04-11 (Actual); Study Completion 2022-04-11 (Actual)

PRIMARY OUTCOMES:
Phase 1 Dose Escalation - Regimens A, B,and C: Incidence of dose limiting toxicities (DLTs) | Regimen A and B dose escalation Days 1-21, Regimen C dose escalation Days 8-36 days
Phase 1 Dose Escalation - Regimens A, B, and C and Phase 1 Expansion - Regimen B: Incidence of adverse events (AEs) | Regimen A and C from first dose through 30 days post last dose, Regimen B from first dose through 90 days post last dose
Phase 1 Dose Escalation - Regimens A and B: Cmax of GB1275 | From first dose through 30 days post last dose
  Maximum observed plasma concentration
Phase 1 Dose Escalation - Regimens A and B: Ctrough of GB1275 | From first dose through 30 days post last dose
  Trough observed plasma concentration
Phase 1 Dose Escalation - Regimens A and B: Tmax of GB1275 | From first dose through 30 days post last dose
  Time of maximum observed plasma concentration
Phase 1 Dose Escalation - Regimens A and B: t1/2 of GB1275 | From first dose through 30 days post last dose
  Terminal phase elimination half-life
Phase 1 Dose Escalation - Regimens A and B: AUC of GB1275 | From first dose through 30 days post last dose
  Area under the plasma concentration-time curve
Phase 1 Dose Escalation - Regimens A and B: CL/F of GB1275 | From first dose through 30 days post last dose
  Oral clearance
Phase 2 - Basket Cohorts 1, 2 and 3: Objective Response Rate (ORR) | 24 months
  ORR defined as the proportion of subjects with best overall confirmed response (BOCR) of either a complete response (CR) or partial response (PR) as assessed by the Investigator based on RECIST v1.1

SECONDARY OUTCOMES:
Phase 1 - Regimen C and Phase 1 Expansion - Regimen B: Cmax of GB1275 | From first dose through 30 days post last dose
  Maximum observed plasma concentration
Phase 1 - Regimen C and Phase 1 Expansion - Regimen B: Ctrough of GB1275 | From first dose through 30 days post last dose
  Trough observed plasma concentration
Phase 1 - Regimen C and Phase 1 Expansion - Regimen B: Tmax of GB1275 | From first dose through 30 days post last dose
  Time of maximum observed plasma concentration
Phase 1 - Regimen C and Phase 1 Expansion - Regimen B: t1/2 of GB1275 | From first dose through 30 days post last dose
  Terminal phase elimination half-life
Phase 1 - Regimen C and Phase 1 Expansion - Regimen B: AUC of GB1275 | From first dose through 30 days post last dose
  Area under the plasma concentration-time curve
Phase 1 - Regimen C and Phase 1 Expansion - Regimen B: CL/F of GB1275 | From first dose through 30 days post last dose
  Oral clearance
Phase 1 - Regimen C: Cmax of nab-paclitaxel and gemcitabine | From first dose through 30 days post last dose
  Maximum observed plasma concentration
Phase 1 - Regimen C: Tmax of nab-paclitaxel and gemcitabine) | From first dose through 30 days post last dose
  Time of maximum observed plasma concentration
Phase 1 - Regimen C: AUC of nab-paclitaxel and gemcitabine | From first dose through 30 days post last dose
  Area under the plasma concentration-time curve
Phase 2 - Basket Cohorts 1, 2, and 3: Duration of Response (DOR) | 24 months
  DOR defined as time from date of objective response to first documented date of disease progression or death
Phase 2 - Basket Cohorts 1, 2, and 3: Time to Response (TTR) | 24 months
  TTR defined as time from first dose to first date of objective response
Phase 2 - Basket Cohorts 1, 2, and 3: Clinical Benefit Rate (CBR) | 6 months
  CBR defined as proportion of subjects with confirmed CR, PR, or stable disease (SD) at six months.
Phase 2 - Basket Cohorts 1, 2, and 3: Progression Free Survival (PFS) | 24 months
  PFS defined as time from first dose to first documented date of disease progression or death.
Phase 2 - Basket Cohorts 1, 2, and 3: Time to Progression (TTP) | 24 months
  TTP defined as time from first dose to first documented date of disease progression.
Phase 2 - Basket Cohorts 1, 2, and 3: Overall Survival (OS) | 24 months
  OS defined as time from first dose to date of death.
Phase 2 - Basket Cohorts 1, 2, and 3: Incidence of AEs | Basket Cohorts 1 from first dose through 30 days post last dose, Basket Cohorts 2 and 3 from first dose through 90 days post last dose.
Phase 2 - Basket Cohort 1, 2 and 3: PK profile of GB1275 | Basket Cohorts 1, 2, and 3 from first dose through 30 days post last dose.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (7):
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - University of Colorado Hospital, Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Sarah Cannon Research Institute/Tennessee Oncology, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- The Royals Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No